CLINICAL TRIAL: NCT06518668
Title: A Phase 1 Study of NKX019, a CD19 Chimeric Antigen Receptor Natural Killer (CAR NK) Cell Therapy, in Subjects With Systemic Lupus Erythematosus
Brief Title: A Study of NKX019, a CD19 CAR NK Cell Therapy, in Subjects With Systemic Lupus Erythematosus
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Columbia University (Other)
Responsible Party: Principal Investigator, Anca Askanase, Professor of Medicine, Columbia University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AAAV0505
Record Dates: First submitted 2024-07-19; First posted 2024-07-24 (Actual); Last update posted 2025-07-25 (Actual); Status verified 2025-07

CONDITIONS: Systemic Lupus Erythematosus
Keywords: CD19; CAR; Allogeneic; NKX019; Cell Therapy; Lupus Nephritis; Systemic lupus erythematosus
MeSH Terms: conditions — Lupus Erythematosus, Systemic; Lupus Nephritis | interventions — Cyclophosphamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- NKX019 infusion (Experimental): Subjects with SLE will receive cyclophosphamide LD followed by NKX019.
  Interventions: Biological: NKX019; Drug: Cyclophosphamide LD

INTERVENTIONS:
Biological: NKX019 — NKX019 is an investigational allogeneic CD19-Directed CAR NK. NKX019 will be administered at a dose of 1 × 109 CAR NK cells (dose normalized for weight for subjects ≤ 50 kg) administered IV.
  Other Names: NKX019 infusion
Drug: Cyclophosphamide LD — Cy dose of 1 g/m2 administered IV over 30 to 60 minutes for the purpose of Lymphodepletion Therapy. Cyclophosphamide will help prepare your body to receive the treatment by decreasing the cells from your immune system to make space for the NKX019 cells.
  (non-experimental)
  Other Names: Cy

SUMMARY:
Primary objective: Safety and tolerability of NKX019, administered after lymphodepletion (LD).

Secondary objectives:

* Assess clinical activity of NKX019 in subjects with systemic lupus erythematosus (SLE) with or without active lupus nephritis (LN)
* Characterize pharmacokinetics (PK) of NKX019
* Characterize immunogenicity of NKX019

DETAILED DESCRIPTION:
This is an open-label, non-randomized, Phase 1 study. Subjects with SLE will receive cyclophosphamide LD followed by NKX019 to determine safety and preliminary efficacy.

The study will consist of 4 study periods for each study subject inclusive of Screening, Active Treatment, Follow-up, and Extended Follow-up. Disease assessments will occur every 90 days for 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18-65 years old at the time of informed consent
* Signed informed consent form, able to adhere to the study visit schedule, and comply with other requirements of the study as specified in the protocol
* Score of 8 or more points on the Hybrid-SLEDAI with at least 6 points from clinical items and at least one BILAG A or 2 B
* If SLE and LN: Active nephritis Class III or IV with or without Class V using the 2018 International Society of Nephrology and Renal Pathology Society (ISN/RPS) criteria as evidenced on kidney biopsy during screening or within 12 months before study enrollment. Per NIH indices, subjects must have at least activity score ≥ 2 and no more than moderate chronicity index. Subjects must have urinary protein:creatinine ratio (UPCR) ≥ 1.5 g/g or proteinuria ≥ 1.5 g/day, however, subjects must have ≤7g/ day of proteinuria.
* For patients with biopsies older than 6 months we will include an adjudication committee to review clinical data and decide on appropriateness of including the patient (see section 7.3). Additionally, all patients with active LN maximally tolerated doses of renin angiotensin aldosterone system (RAAS) blockade agents, except for patients with contraindications or intolerance to RAAS.
* Women of childbearing potential must have a negative serum pregnancy test at screening and agree to complete abstinence from intercourse from 2 weeks prior to administration of the first dose of study agent until 1 year after the last dose of study agents OR consistent and correct use of acceptable birth control (e.g. levonorgestrel implants, ethinyl estradiol/etonogestrel vaginal ring; injectable progesterone, intrauterine device [IUD] with failure rate < 1% per year, oral contraceptives, double barrier method, transdermal contraceptive patch) OR male partner sterilization with documentation of azoospermia prior to subject's entry into the study.
* Male patients must agree to always use a latex or other synthetic condom during any sexual activity with women of childbearing potential. Male participants must agree to continue to use a condom during the intervention period and for at least 1 year following last treatment with investigational product. Female partners of male participants should be advised to use a highly effective method of contraception during treatment period and at least 12 months following treatment.
* One of the following: positive antinuclear antibodies (ANA) ≥ 1:80 at screening OR positive anti-dsDNA OR positive anti-Smith (anti-Sm) as determined by the local laboratory.
* Refractory SLE defined as having received ≥ 2 prior therapies for SLE (one immunosuppressant and one biologic/advanced therapy) and had an inadequate response to therapy despite being on a therapeutic dose for ≥ 90 days.
* For subjects taking chronic corticosteroids for SLE/LN management, the dose must be stable for ≥ 14 days before screening and cannot exceed 20 mg prednisone/day or equivalent at LD start with planned taper to ≤ 5 mg prednisone by the time of LD start with planned taper to ≤ 5 mg prednisone by the time of the first NKX019 infusion.
* Negative SARS-CoV-2 test.

Exclusion Criteria:

* Estimated glomerular filtration rate (eGFR) as calculated by the Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) equation of < 45 mL/min/1.73 m2 at screening.
* Currently requiring renal dialysis (hemodialysis or peritoneal dialysis) or expected to require dialysis during the study period
* More than 7 g/ day of proteinuria.
* Previous solid organ or hematopoietic cell transplant or planned transplant within study treatment period.
* Congenital or acquired immunodeficiency resulting in severe infection or those receiving chronic immunoglobulin replacement therapy.
* Liver disease or dysfunction, including cirrhosis and/or aspartate aminotransferase, alanine aminotransferase, or bilirubin ≥ 3 times the upper limit of normal.
* Pulmonary comorbidity including chronic obstructive pulmonary disease or asthma requiring daily oral steroids or resting hypoxemia (< 90% oxygen saturation via pulse oximetry) on room air.
* >10 pack years of smoking.
* Exacerbation of COPD/asthma requiring systemic steroid therapy within the past 6 months.
* Bone marrow insufficiency unrelated to active SLE (according to Investigator judgment) with white blood cell count < 1,500/mm3; hemoglobin levels < 9 g/dL absolute neutrophil count (ANC) < 1,000/mm3; absolute lymphocyte count </=500 mm3, or platelet count ≤ 75,000/mm3
* Major cardiac disease, abnormalities, or interventions as defined by, but not limited to:

  1. Uncontrolled angina or unstable life-threatening arrhythmias
  2. History of myocardial infarction within 12 weeks prior to the first dose of NKX019
  3. Any prior coronary artery bypass graft surgery
  4. ≥ Class III New York Heart Association (NYHA) congestive heart failure (CHF), significantly decreased ejection fraction (EF ≤ 45%), or severe cardiac insufficiency
  5. Prolongation of the QT interval corrected for heart rate (QTc) (Fridericia) interval of > 480 msec
  6. Peripheral artery bypass graft surgery, pulmonary embolism, or other ≥ Grade 2 thrombotic or embolic events within 12 weeks prior to the first dose of NKX019 12. Active CNS SLE . 13. Active bleeding disorders.
* Any overlapping autoimmune condition for which the condition or the treatment of the condition may affect the study assessments or outcomes (e.g. scleroderma with significant pulmonary hypertension; any condition for which additional immunosuppression is indicated). Overlapping conditions for which the condition or treatment is not expected to affect assessments or outcomes (e.g. Sjögren's syndrome) are not excluded.
* Pregnancy, breast feeding or, if of childbearing potential, not using adequate contraceptive precautions or planned oocyte and sperm donation.
* Current/active infection, and any infection requiring systemic antimicrobial therapy within the past 30 days of planned LD.
* History of positive HIV antibody or test positive at screening. Hepatitis B or C positive at screening, active tuberculosis (TB) or latent TB requiring suppressive therapy.
* Major surgery within 28 days prior to the first dose of NKX019 or any surgery from which the subject has not recovered or has ongoing complications.
* Malignancy within 5 years of screening, with the exception of basal and squamous cell carcinomas treated by complete excision. Subjects with cervical dysplasia that is cervical intraepithelial neoplasia but have been treated with conization or loop electrosurgical excision procedure, and have had a normal repeat Papanicolaou test are allowed.
* Prior cellular therapy, including mesenchymal, CAR-T or CAR-NK cells.
* Prior cerebrovascular ischemia/hemorrhage including transient ischemic attack within 90 days prior to the first dose of NKX019.
* Any other acute or chronic medical or psychiatric condition, or known laboratory abnormality that, in the Investigator's opinion is expected to:

  1. Increase the risk associated with study participation or NKX019 administration
  2. Interfere with the informed consent process, compliance with the study requirements, or interpretation of the study results
  3. Make the subject inappropriate for entry into this study
  4. Require concomitant use of any medication that is listed as prohibited while on study
  5. In the opinion of the Investigator, clinically significant drug or alcohol abuse within 2 years prior to screening
* Prior therapies for SLE, including investigational agents, within 4 weeks or 5 half-lives of the drug (whichever is longer) prior to lymphodepletion.
* Currently taking or known need for any of the medications prohibited in the study protocol.
* Known hypersensitivity or contraindications to the study treatment including LD; or other components such as human serum albumin or dimethyl sulfoxide.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Estimated)
Dates: Start 2024-07-01 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2040-12 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse events (AEs) | 2 years
  This is to measure safety and tolerability of NKX019, administered after lymphodepletion (LD). Adverse events will be graded using National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) v5.0, including dose-limiting toxicities (DLTs). A DLT is defined as an AE or clinically significant laboratory abnormality (laboratory abnormalities, including transient [lasting < 24 hours] or isolated out of range values) occurring within 28 days from the first dose that is possibly attributable to NKX019.

SECONDARY OUTCOMES:
Change from baseline of autoantibody levels | Up to 2 years after NKX019 infusion
  This is to measure/assess clinical activity of NKX019 in subjects with systemic lupus erythematosus (SLE) with or without active lupus nephritis (LN). Anti-double-stranded DNA (anti-dsDNA) antibodies and complement levels will be assessed at Days 90, 180, 270, and 360. Change will be evaluated from baseline of autoantibody and complement assessment as follows: Autoantibodies and Complement (C3, C4) levels.
Change from baseline in hybrid SLEDAI (Systemic Lupus Erythematosus Disease Activity Index) score | Up to 2 years after NKX019 infusion
  This to measure/assess clinical activity of NKX019 in subjects with systemic lupus erythematosus (SLE) with or without active lupus nephritis (LN). SLEDAI score (obtained by adding the individual 24 item scores) ranges from 0 to 105, where the higher the score, the greater the degree of disease activity. Score of 6 or more are consistent with therapy requirement.
Number of participants who achieved renal response | Up to 2 years after NKX019 infusion
  This to measure/assess clinical activity of NKX019. For subjects with LN: Assess complete renal response (CRR) and partial renal response (PRR) per European Alliance of Associations for Rheumatology (EULAR)/European Renal Association-European Dialysis and Transplantation Association (ERA-EDTA) criteria.
Maximum concentration (Cmax) of PK in peripheral blood | Up to 2 years after NKX019 infusion
  This is to characterize pharmacokinetics (PK) of NKX019 and evaluate PK parameters.
Number of subjects with normalized serological activity | Up to 2 years after NKX019 infusion
  This is to characterize immunogenicity of NKX019 and assess humoral and cellular immunogenicity over time. Subjects will be followed at 12 weeks and overtime for normalized serological activity such as:
  * Autoantibodies (anti-dsDNA, ANA, and anti-Sm) present to absent
  * Complement (C3, C4, and C3 AND C4) levels low to normal/high

CONTACTS AND LOCATIONS:
Overall Officials: Anca D Askanase, MD, MPH, Principal Investigator — Columbia University
Locations (1):
- Columbia University Irving Medical Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No